CLINICAL TRIAL: NCT02837406
Title: Evaluation of the Implementation and Results of the Health Digital Territories Program in the Five Pilot Territories (EvaTSN Project )
Brief Title: Evaluation of the Health Digital Territories Program in the Five Pilot Territories (EvaTSN Project )
Acronym: EvaTSN
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2014/42
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Evaluation of a National Health Information Technology-based Program to Improve Healthcare Coordination and Access to Information

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Doctors: specialists and general practitioners by ich territory
- Health professionals: * pharmacists
  * nurses
  * physiotherapists
  * Medical and social professionals: social workers, psychologists, educators ...
- Medical-social institutes: * Hospital,
  * Healthcare structure,
  * Local Centre of Information and Gerontological Coordination ...

SUMMARY:
The aim is to evaluate a national health information technology-based program to improve healthcare coordination and access to information.

DETAILED DESCRIPTION:
Improvement of coordination of all health and social care actors in the patient pathways is an important issue in many countries; Health Information (HI) technology has been considered as a potentially effective answer to this issue. The French Health Ministry first funded the development of five TSN ("Territoire de Soins Numérique" / Digital health territories) programs, aiming at improving healthcare coordination and access to information for healthcare providers, patients or the population, and at improving healthcare professionals work organization; The French Health Ministry then launched a call for grant to fund one Eva TSN project consisting in evaluating the TSN programs implementation and impact and to develop a model for HI technology evaluation.

ELIGIBILITY:
* Patients(people living in the five pilot territories of the Health Digital Territories program and the five control territories
* 'Users' who used the devices implemented, including platforms computerized,
* "Health professionals" : which includes both the health professions, medical and social professionals and groups representing them (URPS, etc.) and health facilities
* "Governance bodies" such as Regional Hospitalization Agency, the local authorities, etc.
* Manufacturers responsable for implementation of considered digital solutions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health professionals, primary care physicians (General Practitioner ), other liberal medical professionals, hospital practitioners, field professionals, medical social, users of evaluated systems, patients, industrial responsable of digital health program
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Type and number of services developed for professionals | June 2018

SECONDARY OUTCOMES:
Number of users who are familiar with the program | June 2018
Number of users (professional and / or patient / citizen) | June 2018
Number of clicks by professional and / or user patient / citizen | June 2018
Online time (start, end) by professional and / or user patient / citizen | June 2018
Relevance rate of short stay admissions | june 2018
Rates of preventable hospital stays | June 2018
Rate of irrelevant drug prescriptions | June 2018
Rate of recourse to prevention programs | June 2018

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Rachid SALMI, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - Agences Régionales de Santé Bourgogne, Chalon-sur-Saône
  - Agence régionale de santé de Rhône Alpes, Lyon
  - Agences Régionales de Santé Aquitaine, Mont-de-Marsan
  - Agence Régionale de Santé (ARS) Ile-de-France, Paris
  - Agence Régionale Santé Océan Indien, Saint-Denis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saillour-Glenisson F, Duhamel S, Fourneyron E, Huiart L, Joseph JP, Langlois E, Pincemail S, Ramel V, Renaud T, Roberts T, Sibe M, Thiessard F, Wittwer J, Salmi LR; EvaTSN Research group. Protocole of a controlled before-after evaluation of a national health information technology-based program to improve healthcare coordination and access to information. BMC Health Serv Res. 2017 Apr 21;17(1):297. doi: 10.1186/s12913-017-2199-y. PMID 28431579